CLINICAL TRIAL: NCT05902325
Title: Identifying Predictors Of Long-Lasting Response To Mepolizumab In CRSwNP: Is The Disease-Modifying Role Secondary To Restored Anti-Viral Activity Or Enhanced Epithelial Regeneration?
Brief Title: Identifying Predictors Of Response To Mepolizumab In CRSwNP
Acronym: ISS-RESMEPO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-11343
Record Dates: First submitted 2023-05-11; First posted 2023-06-15 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: CRSwNP; Epigenetic; Virus; Multiomics; Mepolizumab
MeSH Terms: conditions — Virus Diseases | interventions — mepolizumab; Injections

STUDY DESIGN:
Intervention Model Description: Patients with severe recurrent CRSwNP will receive Mepolizumab 100mg SC once every 4 weeks for 48 weeks (twelve injections, no placebo) at the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mepolizumab 100mg injection (Experimental): Mepolizumab 100mg SC once every 4 weeks for 48 weeks (twelve injections)
  Interventions: Drug: Mepolizumab 100 MG Injection

INTERVENTIONS:
Drug: Mepolizumab 100 MG Injection — Patients will receive Mepolizumab 100mg SC once every 4 weeks for 48 weeks (twelve injections, no placebo) at the hospital. The IMP will be administered following clinic procedures and blood collection. Patients will be monitored at the study site for at least 30 minutes after injections for signs of hypersensitivity reaction. Subcutaneous injection sites should be alternated among the 4 quadrants of the abdomen (avoiding navel and waist areas) or the upper arms. Background therapy will be assured with mometasone furoate nasal spray (200µg BID) daily throughout the study.
  Other Names: Nucala

SUMMARY:
The investigators propose a real-world study to assess the mechanism of action of long-lasting response to mepolizumab in patients with chronic rhinosinusitis with nasal polyposis (CRSwNP) and identify clinically useful predictors of response.

Mepolizumab is a monoclonal antibody targeting IL-5 and is approved for use in asthma and CRSwNP. In clinical studies, 12 months of treatment with mepolizumab improved signs and symptoms of CRSwNP and reduced the need for surgery. While several biologic medications targeting facets of the Type 2 mechanism are currently indicated for chronic rhinosinusitis with nasal polyps mepolizumab alone appears capable of modifying the disease's biological behaviour and producing long-standing improvements after the cessation of treatment. In the mepolizumab for CRSwNP regulatory trial (SYNAPSE), a subset of patients experienced dramatic and long-lasting, which is over 48 months after cessation of administration of the investigational medicinal product (IMP) in our experience. This has been partially captured in a follow-on study to the registration trail, which showed that a subset of patients followed for 24 weeks after cessation of biologic therapy (with continued use of mometasone furoate) demonstrated persistent improvements over baseline.

However, the mechanism of the long-lasting effect in a subset of patients is not well understood, and it is impossible currently to identify patients who will derive this maximal benefit. The mechanism for the prolonged improvements in CRSwNP seen in certain patients with mepolizumab remains to be established but suggests that effects beyond eosinophil trafficking are implicated.

The investigators believe that mepolizumab has IL-5-mediated pleiotropic effects which contribute to disease modification with effects extending beyond eosinophil activation and trafficking. This may include the following primary or secondary effects:

i) Improving epithelial barrier function ii) Altering mast cell dynamics iii) Reversing epigenetic modifications iv) Altering the immune response to better clear pathogenic bacteria or viruses.

DETAILED DESCRIPTION:
Study Rationale:

The investigators propose an ambitious research program to investigate the underlying mechanism of action of the prolonged responses to treatment with mepolizumab in patients with CRSwNP seen in the SYNAPSE trial. In addition, the investigators seek to establish the link between viral disease and eosinophilia, based upon a concept of viral interference with immunologic response inspired by findings from the COVID-19 pandemic.

Study Design:

In this monocentric prospective cohort study, two seasoned investigators will assess the disease-modifying effects of mepolizumab on CRSwNP. This study aims to identify in a ''real-world'' setting the mechanisms underpinning the prolonged response to mepolizumab and identify biomarkers predictive of prolonged response. Thirty-six patients with CRSwNP unresponsive to medical and surgical treatment will be treated with twelve months of mepolizumab in an unblinded and nonrandomized fashion (open-label).

The response will be assessed with usual clinical parameters, including sino-nasal endoscopy. The mechanism of response will be explored in depth before and 6 months after the beginning of treatment with a multiomic approach. The long-term effect will be assessed by clinical assessment only.

1. Determine the mechanism of action of mepolizumab in CRSwNP with multiomics. The investigators will explore the critical mechanisms that contribute to transcription patterns in diseased tissue in a cell-type-specific perspective and explore whether viral infection contributes to CRS. Simultaneous profiling of gene expression and open chromatin from the same cell will be used to capture epigenetic modifications in identified cell clusters by RNA-seq combined with an assay for transposase-accessible chromatin (Chromium Single-Cell Multiome ATAC + Gene expression, 10X Genomics).
2. Confirm improved epithelial regeneration and repair following mepolizumab treatment via in vitro functional assessment of epithelial capacity for regeneration.

   Using in vitro wound healing models, the investigators will evaluate the proliferation and cell migration of PEC from patients' nasal polyp biopsy prior to and 6 months after the beginning of treatment. Each time point will be assessed in triplicate on petri (3 wells/ patient) along with cultures on Lab-Tek chamber slides for immunofluorescence assays. Functional assessment of the capacity of tissue repair will be assessed by the speed of repair following standardized injury. Immunofluorescence will assess the markers of the epithelium (tubulin, cadherin, vimentin etc.) and epithelial function (tight junction, zonula occludens, integrins etc.) and by the presence of proliferation markers (Ki-67) at the wound site.
3. Identify associated epigenetic marks of response which can serve as potential biomarkers of the responder population.

   As described above, epigenetic modulation of the genome will be assessed at the single-cell level in multiomic profiling. In order to restrict epigenetic profiling to epigenetic modifications which may have a use as biomarkers, DNA methylation profiling will be performed by DNA MethylationEPIC Beadchip to identify putative biomarkers of response to treatment and identify methylation-related regulatory mechanisms.
4. Characterise the impact of mepolizumab on viruses by defining a library of viruses present in CRSwNP and comparing their levels pre- and post-treatment with mepolizumab.

   The investigators will perform sequenced-based profiling using deep sequencing technologies (Illumina high-throughput RNA sequencing) to reveal candidate viral pathogens using an existing pre-COVID biobank of CRSwNP tissue in our institution to define the type of viruses present in CRSwNP. Similarly, viruses will be assessed in the population undergoing treatment with mepolizumab to assess whether treatment influences viral burden and specific viruses.
5. Identify epigenetic marks associated with the presence of different viruses which can serve as markers of prior viral infection.

The investigators will investigate the specific association between viruses and epigenetic marks with the integrative analysis of the resulting data using epigenomics and transcriptomics methods.

There will be a follow-up of patients over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral NP, as diagnosed by endoscopy or historical CT scan
* At least one NP surgery* within the last 10 years.
* Severe NP symptoms consistent with a need for surgery (obstruction VAS symptom score>5, overall, VAS symptom score >7, endoscopic bilateral NP score ≥4 [with a score ≥2 in each nasal cavity]).
* Ongoing treatment with INCS (via spray or intranasal liquid steroid wash/douching) for ≥4 weeks prior to screening
* ≥2 of the following CRS symptoms for at least 12 weeks:

  * Nasal blockage/obstruction/congestion
  * Nasal discharge (anterior/posterior nasal drip)
  * Facial pain/pressure
  * Reduction or loss of sense of smell

Exclusion Criteria:

* If as a result of a medical interview, physical examination, or screening investigation the physician responsible considers the participant unfit for the study.
* Cystic fibrosis
* Eosinophilic granulomatosis with polyangiitis (also known as Churg Strauss syndrome), Young's, Kartagener's or dyskinetic ciliary syndromes
* Antrochoanal polyps
* Nasal septal deviation occluding one nostril
* Acute sinusitis or upper respiratory tract infection (URTI) at screening or 2 weeks prior to screening
* Ongoing rhinitis medicamentosa (rebound or chemical-induced rhinitis)
* Participants who have undergone any intranasal and/or sinus surgery (for example polypectomy, balloon dilatation or nasal stent insertion) within 6 months prior to V1
* Participants where NP surgery is contraindicated in the opinion of the Investigator
* Participants with a known medical history of HIV infection.
* Participants with a known, pre-existing parasitic infestation within 6 months prior to Visit 1.
* Participants who are currently receiving or have received within 3 months (or 5 half-lives - whatever is the longest) prior to the screening visit, radiotherapy, or investigational medications/therapies.
* Participants with a history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. Aspirin-sensitive participants are acceptable.
* Participants with a history of allergic reaction to anti-IL-5 or other monoclonal antibody therapy.
* Use of systemic corticosteroids (including oral corticosteroids) within 4 weeks prior to screening or planned use of such medications during the double-blind period
* Treatments with biological or immunosuppressive treatment (other than Xolair) treatment within 5 terminal phase half-lives of Visit 1
* Omalizumab (Xolair) treatment in the 130 days prior to Visit 1
* Commencement or change of dose of allergen immunotherapy within the previous 3 months.
* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study. Contraceptive use will be required with a double barrier method or documented effective surgical sterilization.
* Immunocompromised subjects from disease or medication, other than oral corticosteroids.
* Women of childbearing potential (WOCBP) will be included with measures to prevent accidental exposure to IMP by using double barrier contraception and pregnancy test prior to injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Persistent clinical response to mepolizumab after cessation off mepoluzimab treatment | 18 months
  Percentage (%) of participants demonstrating persistent clinical response to mepolizumab following cessation of treatment will be defined as persistence of improvement in Nasal Polyp size greater than 1 six months after cessation of a twelve-month treatment course of mepoluzimab.

OTHER OUTCOMES:
Determine effect of mepolizumab on trafficking of individual immune and structural cell types present in the epithelium in CRSwNP | 6 months
  Single-cell transcriptomic techniques will be used to identify cell types present in CRSwNP biopsy samples. Relative proportion identified cell types will be defined, and compared at pre-treatment and after 6 months of treatment with mepolizumab.
Effect on epithelial function in vitro | 6 months
  In vitro wound repair speed will be measured in primary epithelial cell (PEC) cultures raised from the patients, before and at 6-month time point of mepolizumab treatment.
Effect on epithelial function in vivo | 6 months
  Impact of mepolizumab on In vivo epithelial development and differentiation will be verified by gene expression profiling. Endoscopically-collected epithelial brushings will be collected before and after mepoluzimab treatment. Samples will be processed to undergo expression proofing to assess activity of genes associated with epithelial proliferation and differentiation in Gene Set Ontology (GSEA) Hallmark network.
Identify viruses associated with CRSwNP. | 6 months
  A library of frozen samples biopsies taken from CRSwNP patients undergoing ESS for inflammatory disease will be compared with control subjects undergoing access procedures to the skull base . Viruses will be defined as 'significantly present' if identified in five reads of more of bulk sequencing. Viruses associated with CRSwNP will be defined as those attaining significant levels in tissue (defined as greater than 5 'reads') and not significantly present in healthy tissue.
Explore the modulation of viruses by biological therapy. | 18 months
  Characterize the impact of mepolizumab on viruses by comparing candidate virus levels pre- and post-treatment with mepolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Yvon Desrosiers, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milavetz BI, Balakrishnan L. Viral epigenetics. Methods Mol Biol. 2015;1238:569-96. doi: 10.1007/978-1-4939-1804-1_30. PMID 25421681
- [Background] Jiao J, Wang C, Zhang L. Epithelial physical barrier defects in chronic rhinosinusitis. Expert Rev Clin Immunol. 2019 Jun;15(6):679-688. doi: 10.1080/1744666X.2019.1601556. Epub 2019 Apr 9. PMID 30925220
- [Background] Kim JY, Kim DK, Yu MS, Cha MJ, Yu SL, Kang J. Role of epigenetics in the pathogenesis of chronic rhinosinusitis with nasal polyps. Mol Med Rep. 2018 Jan;17(1):1219-1227. doi: 10.3892/mmr.2017.8001. Epub 2017 Nov 7. PMID 29115522